CLINICAL TRIAL: NCT07069751
Title: A Prospective Multicenter Study of the Effects of Plant-based Diets on Gut Microbiome and Derived Metabolites in Patients Affected by Smoldering Multiple Myeloma
Acronym: HiFi-MM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciceri Fabio (Other)
Responsible Party: Sponsor-Investigator, Ciceri Fabio, MD - Hematology and Bone Marrow Transplant, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HiFi-MM
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Smoldering Multiple Myeloma (SMM)
Keywords: microbiome; plant-based diets; gut microbiome; smoldering multiple myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Enrolled and eligible patients will be encouraged to consume a balanced diet rich in fiber for the entire duration of the trial (i.e., 12 weeks).
  Interventions: Dietary Supplement: diet rich in fiber

INTERVENTIONS:
Dietary Supplement: diet rich in fiber — Enrolled and eligible patients will be encouraged to consume a balanced diet rich in fiber for the entire duration of the trial (i.e., 12 weeks). Patients will also be encouraged to prolong plant-based diets beyond week 12. Free outpatient medical visit will be performed at enrollment and at week 12, and nutritional counseling will be given at the time of enrollment, one month later and on demand. Dietary measurements will be conducted along the entire duration of the nutritional regimen by questionnaires. In particular, the patient will write for each day of the trial the number associated to the chosen diet plan or food.

SUMMARY:
Our overarching hypothesis is that plant-based diets will induce beneficial modifications of the gut microbiota favoring short fatty acid (SCFA)-producing commensals and a more advantageous CD8/Th17 ratio in sMM patients, thus preventing evolution to MM. Goal of this national, prospective, multicenter study is to demonstrate that plant-based diets substantially modify the gut microbiome inducing increased production of SCFAs in patients affected by sMM. The study will involve up to 62 patients affected by sMM. 56 Enrolled and eligible patients will be encouraged to consume a balanced diet rich in fiber for the entire duration of the trial (i.e., 12 weeks). Patients will choose among a list of different diet plans or individual food according to the personal tastes and preference. Free outpatient medical visit will be performed at enrollment and at week 12, and nutritional counseling will be given at the time of enrollment, one month later and on demand. As in line with routine diagnosis and follow-up of for patients affected by sMM, the investigators will collect bone marrow aspirates and peripheral blood at the time of screening, for plasma, serum, and peripheral blood mononuclear cells (PBMCs), while stool samples will be collected immediately before diet initiation. The investigators will also collect stool samples 4 and 12 weeks after diet initiation, and peripheral blood at 12 weeks after study initiation (as per routine clinical follow-up of this patient population). Dietary measurements will be conducted along the entire duration of the nutritional regimen by questionnaires. Biological paired comparison will be conducted between data obtained from samples collected at time 0 and samples collected 4 and 12 weeks later.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent for participation in the study.
2. Confirmed diagnosis of sMM according to IMWG criteria
3. Absence of features of symptomatic or active myeloma requiring treatment (myeloma-defining events).
4. Aged ≥18 and </= 75 years
5. Participant is willing to comply with all study-related procedures.
6. ECOG performance status of 0-1.

Exclusion Criteria:

1. Non-Caucasian subjects. Racial disparities in all stages of the disease characterize MM, and Blacks have an increased MGUS and MM risk and higher mortality rate than Whites.
2. Patients that already follow a whole food plant-based diet (≥ 40g/die;ovo-lacto-vegetarian or processed junk food vegan diets are not excluded). These patients likely should already have high SCFA levels in their gut.
3. Legume allergy.
4. Severe allergies such as anaphylactic shock to nuts (specifically cashews).
5. Concurrent participation in weight loss/dietary/exercise programs because of potential conflicts between the concurrent diet and high-fiber diet.
6. Enrollment onto any other therapeutic investigational study.
7. Concurrent pregnancy.
8. Ongoing treatment for HBV, HCV or HIV.
9. If in the opinion of the investigator there maybe any concerns regarding the ability of the patient to complete the study safely or any contraindications.
10. Heavy drinker (defined as >2 drinks per day or >14 drinks per week).
11. Current self-reported illicit drug use (e.g., heroin, cocaine not marijuana).
12. Subjects that did not accept to sign the informed consent.
13. Subjects reporting infectious diseases requiring antibiotic therapy in the previous three months, ongoing antibiotic therapy, or prophylaxis. Antibiotic therapy dramatically modifies the composition of the gut microbiota.
14. Subjects affected by autoimmune diseases except for thyroiditis, and patients affected by small and large intestine dysfunctions (i.e., inflammatory bowel disease).
15. Gammopathy-associated conditions beyond sMM (e.g. amiloydosis, POEMS, LCDD, etc).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of high-fiber diets on mean SCFA concentration in stool samples. | Stool sampling at day 0, 28 and 84 since high-fiber diet starts.
  Concentration of at least one among the three main SCFAs (acetate, butyrate and propionate) in stool samples from participants.
  Stool samples will be collected at Baseline visit (day 0) and 4 and 12 weeks later.
  SCFAs will be measured by targeted nuclear magnetic resonance.

SECONDARY OUTCOMES:
To evaluate adherence to the diet regimen. | Daily dietary measurement by questionnaires and food diary and dietary interview (30 minutes, either in-presence or virtually) at day 0, 28 and 84 since high-fiber diet starts.
  Frequency of participants adhering to the high-fiber diet (≥ 40g/die) at week 4 and 12 weeks since the start.
To evaluate the effects of high-fiber diets on gut microbiome composition. | Stool sampling at day 0, 28 and 84 since high-fiber diet starts.
  Composition of the gut microbiota. Stool samples will be collected at Baseline visit (day 0) and 4 and 12 weeks later.
  Composition of the gut microbiota will be obtained by 16S ribosomal RNA sequencing of paired stool samples.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale Giovanni XXIII Policlinico di Bari, Bari
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma